CLINICAL TRIAL: NCT02463279
Title: SinuSys Patency of Frontal Recess and Sphenoid Sinus Ostia Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SinuSys Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNS-006
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SinuSys Dilation System (Experimental): Opening of previously constrained frontal recess and/or sphenoid sinus ostia via dilation procedure (sinuplasty)
  Interventions: Device: Sinusys Dilation System

INTERVENTIONS:
Device: Sinusys Dilation System — Dilation of frontal recess and/or sphenoid sinus ostia

SUMMARY:
The goal of this study is to evaluate basic usability and confirm expected safety and effectiveness of SinuSys Dilation System when used to dilate frontal recess and sphenoid sinus ostia in patients with chronic rhinosinusitis.

DETAILED DESCRIPTION:
A multicenter, single arm, prospective study conducted to assess the safety and effectiveness of an osmotically-drive, low-pressure expansion device for dilation of frontal recess and sphenoid sinus ostia in patients with chronic rhinosinusitis (CRS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CRS
* Subject in in need of frontal recess and/or sphenoid sinus dilation

Exclusion Criteria:

* Pregnant or breastfeeding females
* Previous treatment site intervention
* Cystic fibrosis, aspirin sensitivity, steroid dependent asthma, sinonasal tumors, allergic fungal sinusitis, ciliary dysfunction, atrophic nasal mucosa, excessive osteogenesis that might preclude dilation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Patency of treated target site | Patency immediately post device expansion and removal
  Patency assessed by investigator via endoscopic evaluation of the target site

SECONDARY OUTCOMES:
Patency of treated target site | 1 month and 3 months
  Patency assessed by investigator via endoscopic evaluation of the target site
Reports of sinus related adverse events during the 3 months follow-up period | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Hester, MD, Study Director — SinuSys Chief Medical Officer
Locations (3):
- United States (3):
  - Upland ENT, Upland, California
  - Colorado ENT, Denver, Colorado
  - St. Elizabeth Medical Center, Brighton, Massachusetts